CLINICAL TRIAL: NCT00102908
Title: Bisphosphonate Therapy for HIV-Associated Osteopenia
Brief Title: Bisphosphonate Therapy for HIV-Infected Adults With Decreased Bone Mineral Density
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jeannie S. Huang, MD, MPH, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21AI058756-01 (NIH); 1R21AI058756-01 (NIH)
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections; Osteopenia; Osteoporosis
Keywords: Bone Metabolism; Osteopenia; Osteoporosis; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Bone Diseases, Metabolic; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive zoledronate at study entry; their assigned intervention will be given in a 20- to 30-minute infusion on an outpatient basis
  Interventions: Drug: Zoledronate
- 2 (Placebo Comparator): Participants will receive zoledronate placebo at study entry; their assigned intervention will be given in a 20- to 30-minute infusion on an outpatient basis
  Interventions: Drug: Zoledronate placebo

INTERVENTIONS:
Drug: Zoledronate — Zoledronate infusion
  Arms: 1
Drug: Zoledronate placebo — Zoledronate placebo infusion
  Arms: 2

SUMMARY:
Bisphosphonates are a type of drug used to prevent and treat bone loss. The purpose of this study is to determine if zoledronate, an investigational bisphosphonate, can improve bone mineral density (BMD) in HIV-infected adults.

Study hypothesis: Zoledronate will reduce bone resorption in HIV-infected persons with osteopenia.

DETAILED DESCRIPTION:
Decreased BMD and bone loss is estimated to affect up to 67.5% of the HIV-infected population. HIV-associated bone loss may be a result of antiretroviral treatment (ART), but can also be caused by the infection itself. To date, treatment for this bone loss has not been established. Before prescribing drugs to treat bone loss, physicians must take into account patients' already demanding ART schedules and potential nonadherence. This study will evaluate the efficacy of a single IV dose of zoledronate, an investigational bisphosphonate, in treating HIV-associated bone loss.

This study will last 1 year. Participants will be randomly assigned to receive zoledronate or placebo at study entry; their assigned intervention will be given in a 20- to 30-minute infusion on an outpatient basis. There will be 7 study visits: at screening, study entry, Week 2, and Months 3, 6, 9, and 12. Blood collection will occur at all visits. Medical history, a physical exam, a dual-energy x-ray absorptiometry (DEXA) scan to measure bone density, and a nutrition evaluation will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* On stable antiretroviral regimen for at least 3 months
* Able to walk
* Lumbar spine or total hip BMD T-score at least 1.5 SD and no more than 3.5 SD below the mean BMD
* No prevalent fractures at entry OR 1 prevalent vertebral fracture that has been asymptomatic during the last 2 years prior to study entry
* HIV viral load of less than 5000 copies/ml within the 2 months prior to study entry
* CD4 count of more than 100 cells/mm3 within the 2 months prior to study entry
* Willing to use acceptable forms of contraception during the study period and for 6 months after study completion. Participants who are female and postmenopausal will be required to take hormone replacement therapy during this study.

Exclusion Criteria:

* Prior treatment with bisphosphonates or fluoride
* Use of supraphysiologic systemic estrogen/androgen therapy or corticosteroid therapy within the 3 months prior to study entry. Participants who have taken hormone replacement therapy are not excluded.
* Significant liver or kidney disease
* Hemoglobin less than 8 g/dL
* Serum calcium less than 8 mg/dL
* Laboratory evidence of low levels of estrogens or androgens
* Laboratory evidence of overactive parathyroid glands
* History of thyroid, parathyroid, or other endocrinologic disorder known to affect bone
* Current use of any therapy known to affect bone
* Current or history of cancer or chemotherapy
* Current or history of radiotherapy to the jaw
* Current osteomyelitis of the jaw or ongoing dental infection
* Recent tooth extraction or major dental procedure within 3 weeks of study entry
* Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Bone metabolic markers | Throughout study

SECONDARY OUTCOMES:
Safety outcomes | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie S. Huang, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States